CLINICAL TRIAL: NCT04749875
Title: Study of Leukocyte Populations in Patients With Chronic Inflammatory
Acronym: LIMA
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210093
Record Dates: First submitted 2021-02-06; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Systemic Autoimmune Disease; Chronic Inflammatory Rheumatism; Sjogren's Syndrome; Spondyloarthritis; Rheumatoid Arthritis; Systemic Lupus Erythematosus
Keywords: leukocytes; macrophages; lymphocytes; rare systemic autoimmune diseases; chronic inflammatory rheumatism
MeSH Terms: conditions — Sjogren's Syndrome; Spondylarthritis; Arthritis, Rheumatoid; Lupus Erythematosus, Systemic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sample — sampling of blood for research during routine care

SUMMARY:
Exploration of pathophysiological mechanisms in chronic inflammatory rheumatism and rare systemic autoimmune diseases with the objective of identifying therapeutic targets.

DETAILED DESCRIPTION:
The primary objective is to characterization of the quantitative and qualitative specificities of the different leukocyte sub-populations in patients with chronic inflammatory rheumatism and rare systemic autoimmune diseases. We will perform an exploratory descriptive study whom primary endpoint will be to assess by FACS the phenotype of the specific leukocyte subsets. In addition, we will characterize the protein and transcriptomic signature associated with the conditions for which we have obtained preliminary data showing their potential involvement in autoimmunity (i.e: IL7 pathway, IFN signature).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patient who did not express his opposition
* Patients with chronic inflammatory rheumatism and rare systemic autoimmune diseases (pSS, lupus, scleroderma, myositis, unclassified connectivitis) diagnosed according to the usual criteria.
* Weight> 35 kg

Exclusion Criteria:

* Corticosteroid treatment> 10 mg / day
* Pregnant patient
* Patients under legal protection
* Beneficiary of the state medical aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic inflammatory rheumatism and rare systemic autoimmune diseases
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of the quantitative and qualitative specificities of the different leukocyte subpopulations in patients with chronic inflammatory rheumatism and rare systemic autoimmune diseases | At the end of the study (5 years)
  Proportion of different leukocytes subset

SECONDARY OUTCOMES:
Protein study (ELISA on serum) : IL7 | At the end of the study (5 years)
  levels of IL7 and other cytokines
Transcriptome study (RNA) : mRNA levels | At the end of the study (5 years)
  assessement of different mRRNA involved in Il7/IFN pathways by molecular biology techniques (RNAseq, qPCR, nano string)
Genomic study (DNA) : SNPs | At the end of the study (5 years)
  Determination of the genotype of different SNPs involved in IL7/IFN pathways

CONTACTS AND LOCATIONS:
Overall Officials: Gaetane Nocturne, Principal Investigator — APHP
Locations (1):
- CHU Bicêtre, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No